CLINICAL TRIAL: NCT04867915
Title: Observational Study on the Diagnosis and Management of Chronic Lymphocytic Leukemia (CLL) in Italy by Gruppo Italiano Malattie EMatologiche Dell'Adulto (GIMEMA)
Brief Title: Study on the Diagnosis and Management of CLL in Italy by GIMEMA
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CLL2121
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; MBL-CLL - Monoclonal B-Cell Lymphocytosis Chronic Lymphocytic Leukaemia-Type
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
retrospective and prospective multicenter observational clinical and biological data collection from all patients with newly diagnosed CLL, SLL or MBL.

retrospective cohort: all cases with a diagnosis between January 1st 2010 and August 31th 2021.

prospective cohort: all patients with a diagnosis between September 1st 2021 and September 1st 2025.

DETAILED DESCRIPTION:
This is a retrospective and prospective multicenter observational study designed by the Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA). The study consists of clinical and biological data collection from all patients with newly diagnosed CLL, SLL or MBL (according to the WHO 2007 and 2018 diagnostic criteria). The retrospective part aims at including all cases followed at participating centers with a diagnosis between January 1st 2010 and August 31th 2021 (planned study initiation), while the prospective part will include all patients with a documented diagnosis of CLL, SLL or MBL between September 1st 2021 and September 1st 2025 by the first immunophenotypic/histological evaluation. The data is collected through electronic case report form accessible by the participating centers on a dedicated platform.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at diagnosis
2. One of the following diagnoses that meet the international diagnostic criteria (iwCLL2018 and WHO2017)

   1. Chronic lymphocytic leukemia (CLL)
   2. Small lymphocytic lymphoma (SLL)
   3. CLL-like monoclonal B-cell lymphocytosis (MBL)
3. Retrospective cohort: CLL/SLL/MBL diagnosis between January 1st 2010 and August 31th 2021.
4. Prospective cohort: CLL/SLL/MBL diagnosis between September 1st 2021 and September 1st, 2025.
5. Signed written informed consent according to ICH/EU/GCP and national local laws (if applicable)

Exclusion Criteria:

* - -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with CLL/SLL or MBL diagnosis followed at participant sites starting from January 1st, 2010 (retrospective cohort) and from September 1st, 2021 (prospective cohort).
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Describe the diagnosis and management of CLL patients | at 1 year for the prospective cohort and at 4 years for the retrospective cohort
  evaluation of CLL management in terms of time to first treatment

CONTACTS AND LOCATIONS:
Locations (24):
- Italy (24):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Asst Degli Spedali Civili Di Brescia - Ssvd Centro Trapianti Midollo Per Adulti - Cattedra Di Ematologia, Brescia
  - Asl Brindisi, Ospedale 'Perrino' - Brindisi - Uo Ematologia, Brindisi
  - Fondazione Del Piemonte Per L'Oncologia Centro Trapianti, Candiolo
  - SOD ematologia AOU Careggi, Florence
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - UOC Ematologia AOU Policlinico "G. Martino", Messina
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Ospedale San Raffaele, Milan
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - UOSD Ematologia Giovanni Paolo II, Ragusa
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Ao S. Maria - Terni - Sc Onco Ematologia, Terni
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Asl to 2, Torino Nord Emergenza San Giovanni Bosco - Ssd Ematologia, Torino
  - UOC Ematologia PO Treviso, Treviso
  - UCO Ematologia ASUGI Trieste, Trieste
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza